CLINICAL TRIAL: NCT04607772
Title: A Multicenter, Phase 1/2 Study of Selinexor in Combination With Backbone Treatments or Novel Therapies in Patients With Relapsed or Refractory (RR) Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Study of Selinexor in Combination With Backbone Treatments or Novel Therapies In Participants With Relapsed or Refractory (RR) Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-DLBCL-025
Record Dates: First submitted 2020-10-26; First posted 2020-10-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Keywords: Karyopharm; Diffuse Large B-Cell Lymphoma; DLBCL; KPT-330; Selinexor; Bendamustine; Rituximab; Polatuzumab Vedotin; Gemcitabine; Oxaliplatin; Ibrutinib; Lenalidomide; Tafasitamab; Venetoclax
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — selinexor; Rituximab; Bendamustine Hydrochloride; polatuzumab vedotin; ibrutinib; Lenalidomide; tafasitamab; venetoclax; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm A: Selinexor with Bendamustine and Rituximab (S-BR)) (Experimental): Participants will receive a dose of 40 or 60 or 80 milligrams (mg) of selinexor oral tablets on Days 1, 3, and 8 for Cycle 1 to 6 (each cycle consists of 21 days) during primary treatment and 60 mg on Days 1, 8, 15, and 22 during continuous treatment (each cycle consists of 28 days). Participants will also receive an intravenous (IV) dose of bendamustine 90 milligram per square meter (mg/m^2) on Days 1 and 2 and IV dose of rituximab 375 mg/m^2 on Day 1 during primary treatment for Cycle 1 to 6.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Bendamustine
- Arm B: Selinexor with Polatuzumab Vedotin and Rituximab (S-PR) (Experimental): Participants will receive a dose of 40 or 60 or 80 mg of selinexor oral tablets on Days 1, 3, and 8 for Cycle 1 to 6 (each cycle consists of 21 days) during primary treatment and 60 mg on Days 1, 8, 15, and 22 during continuous treatment (each cycle consists of 28 days). Participants will also receive an IV dose of polatuzumab vedotin 1.8 milligram per kilogram (mg/kg) and IV dose of rituximab 375 mg/m^2 on Day 1 during primary treatment for Cycle 1 to 6.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Polatuzumab Vedotin
- Arm C: Selinexor, Polatuzumab Vedotin, Bendamustine, Rituximab (S-PBR) (Experimental): Participants will receive a dose of 40 or 60 or 80 mg of selinexor oral tablets on Days 1, 3, and 8 for Cycle 1 to 6 (each cycle consists of 21 days) during primary treatment and 60 mg on Days 1, 8, 15, and 22 during continuous treatment (each cycle consists of 28 days). Participants will also receive an IV dose of polatuzumab vedotin 1.8 mg/kg and IV dose of rituximab 375 mg/m^2 on Day 1, and IV dose of bendamustine 90 mg/m^2 on Days 1 and 2 during primary treatment for Cycle 1 to 6.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Bendamustine; Drug: Polatuzumab Vedotin
- Arm D: Selinexor, Rituximab, Gemcitabine, Oxaliplatin (S-R-GemOx) (Experimental): Participants will receive a dose of 40 or 60 or 80 mg of selinexor oral tablets on Days 1 and 3 for Cycle 1 to 6 (each cycle consists of 14 days) during primary treatment and 60 mg on Days 1, 8, 15, and 22 during continuous treatment (each cycle consists of 28 days). Participants will also receive an IV dose of rituximab 375 mg/m^2, IV dose of gemcitabine 1000 mg/m^2, and Oxaliplatin IV dose of 100 mg/m^2 on Day 1 during primary treatment for Cycle 1 to 6.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- Arm E: Selinexor with Ibrutinib and Rituximab (S-IR) (Experimental): Participants will receive a dose of 40 or 60 or 80 mg of selinexor oral tablets on Days 1, 8, and 15 for Cycle 1 to 6 during primary treatment and 40 mg (dose level 1) then 60 mg (dose level 2-4) during continuous treatment (each cycle consists of 28 days). Participants will also receive an IV dose of rituximab 375 mg/m^2 on Day 1, and ibrutinib oral dose of 420 or 560 mg once daily on Day 1 to 28 during primary treatment for Cycle 1 to 6. Participants will also receive ibrutinib oral dose of 420 mg once daily at all dose levels during continuous treatment.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Ibrutinib
- Arm F: Selinexor with Lenalidomide and Rituximab (S-LR) (Experimental): Participants will receive a dose of 40 or 60 mg of selinexor oral tablets on Days 1, 8, and 15 for Cycle 1 to 6 during primary treatment and 40 mg (dose level 1) then 60 mg (dose level 2) during continuous treatment (each cycle consists of 28 days). Participants will also receive an IV dose of rituximab 375 mg/m^2 on Day 1, and lenalidomide oral dose of 20 mg once daily on Days 1 to 21 during primary treatment for Cycle 1 to 6. Participants will also receive lenalidomide oral dose of 20 mg on Days 1 to 21 at all dose levels during the continuous treatment.
  Interventions: Drug: Selinexor; Drug: Rituximab; Drug: Lenalidomide
- Arm G: Selinexor with Lenalidomide and Tafasitamab (S-LT) (Experimental): Participants will receive a dose of 40 or 60 mg of selinexor oral tablets on Days 1, 8, and 15 for Cycle 1 to 12 during primary treatment and 40 (dose level 1) then 60 mg (dose level 2) during continuous treatment (each cycle consists of 28 days). During the primary treatment, participants will also receive lenalidomide oral dose of 25 mg once daily on Days 1 to 21, and tafasitamab IV dose of 12 mg/kg on Days 1, 8, 15, and 22 for Cycle 1 to 3 and Days 1 and 15 for Cycle 4 to 12. Participants will also receive an IV dose of tafasitamab 12 mg/kg on Days 1 and 15 for all dose levels during the continuous treatment.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Tafasitamab
- Arm H: Selinexor with Venetoclax (S-V) (Experimental): Participants will receive 40 or 60 or 80 mg of selinexor oral tablets on Days 1, 8 and 15 for Cycle 1 to 6 of primary treatment and 40 mg (dose level 1) then 60 mg (dose level 2-5) during continuous treatment (28 days per cycle). Participants who received 40 and 60 mg of selinexor during primary treatment will also receive oral dose of venetoclax 200 mg on Days 1 to 7 then 400 mg on Days 8 to 28 for Cycle 1; 400 mg daily for Cycle 2 to 6. Participants who received 60 and 80 mg of selinexor during primary treatment will also receive venetoclax 400 mg orally on Days 1 to 7 then 600 mg on Days 8 to 28 for Cycle 1; 600 mg daily for Cycle 2 to 6. Participants who received 80 mg selinexor during primary treatment will also receive venetoclax 400 mg orally on Days 1 to 7, then 600 mg from Days 8 to 14, then 800 mg from Day 15 to 28 for Cycle 1; 800 mg daily for Cycle 2 to 6. Participants during continuous treatment will also receive venetoclax 400 mg orally daily.
  Interventions: Drug: Selinexor; Drug: Venetoclax

INTERVENTIONS:
Drug: Selinexor — Dose: 40 mg (2 tablets of 20 mg), 60 mg (3 tablets of 20 mg), 80 mg (4 tablets of 20 mg)
  Other Names: KPT-330
Drug: Rituximab — Dose: 375 mg/m^2
  Arms: Arm A: Selinexor with Bendamustine and Rituximab (S-BR)); Arm B: Selinexor with Polatuzumab Vedotin and Rituximab (S-PR); Arm C: Selinexor, Polatuzumab Vedotin, Bendamustine, Rituximab (S-PBR); Arm D: Selinexor, Rituximab, Gemcitabine, Oxaliplatin (S-R-GemOx); Arm E: Selinexor with Ibrutinib and Rituximab (S-IR); Arm F: Selinexor with Lenalidomide and Rituximab (S-LR)
Drug: Bendamustine — Dose: 90 mg/m^2
  Arms: Arm A: Selinexor with Bendamustine and Rituximab (S-BR)); Arm C: Selinexor, Polatuzumab Vedotin, Bendamustine, Rituximab (S-PBR)
Drug: Polatuzumab Vedotin — Dose: 1.8 mg/kg
  Arms: Arm B: Selinexor with Polatuzumab Vedotin and Rituximab (S-PR); Arm C: Selinexor, Polatuzumab Vedotin, Bendamustine, Rituximab (S-PBR)
Drug: Ibrutinib — Dose: 420, 560 mg
  Arms: Arm E: Selinexor with Ibrutinib and Rituximab (S-IR)
Drug: Lenalidomide — Dose: 20, 25 mg
  Arms: Arm F: Selinexor with Lenalidomide and Rituximab (S-LR); Arm G: Selinexor with Lenalidomide and Tafasitamab (S-LT)
Drug: Tafasitamab — Dose: 12 mg/kg
  Arms: Arm G: Selinexor with Lenalidomide and Tafasitamab (S-LT)
Drug: Venetoclax — Dose: 200, 400, 600, 800 mg
  Arms: Arm H: Selinexor with Venetoclax (S-V)
Drug: Gemcitabine — Dose: 1000 mg/m^2
  Arms: Arm D: Selinexor, Rituximab, Gemcitabine, Oxaliplatin (S-R-GemOx)
Drug: Oxaliplatin — Dose: 100 mg/m^2
  Arms: Arm D: Selinexor, Rituximab, Gemcitabine, Oxaliplatin (S-R-GemOx)

SUMMARY:
This is a Phase 1/2, multicenter, open-label study to evaluate the efficacy, and safety of various combinations with selinexor in participants with RR DLBCL. The study will be conducted in two phases: Phase 1 and 2. The Phase 1 of the study will be a standard 3 + 3 dose escalation to determine the maximal tolerated dose (MTD), recommended Phase 2 dose (RP2D) for each treatment arm, and assess the dose limiting toxicities (DLTs). The Phase 2 of the study will be a dose expansion study to assess the efficacy and safety of for RP2D selected at the end of Phase 1 of the study for each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Participants greater than or equal to (≥) 18 years of age.
2. Have pathologically confirmed relapsed/refractory (RR) DLBCL, not otherwise specified (NOS).
3. Participants with High Grade B-cell Lymphoma (HGBL) are allowed in Phase 2 only.
4. Prior lines of systemic therapy for the treatment of DLBCL:

   * For Arms A, B, C, E, F, G, H: Participants must have received at least 1 but no more than 3 prior lines of systemic therapy for the treatment of DLBCL.
   * For Arm D (S-R-GemOx) participants must have received at least 1 but not more than 2 lines of systemic therapy.
5. Positron emission tomography (PET) positive measurable disease per the Lugano Classification 2014, having at least 1 node with longest diameter (LDi) greater than (>) 1.5 centimetres (cm) or 1 extranodal lesion with LDi >1 cm.
6. Adequate bone marrow function at Screening.
7. Circulating lymphocytes less than or equal to (≤) 50 * 109/L.
8. Adequate liver and kidney function.
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
10. An estimated life expectancy of >6 months at Screening.
11. Participants with primary refractory disease defined as no response or relapse within 6 months after ending first-line treatment will be allowed on study (up to 20 percentage [%] of enrolled participants in each Phase).
12. Male participants, and female participants of childbearing potential must agree to use highly effective methods of contraception during the duration of the study and will continue following the last dose of study treatment for the longest duration stated on the label of each of the given drugs (depending on each arm).
13. Female participants of childbearing potential must have a negative serum pregnancy test at Screening. Female participants of childbearing potential in the S-LR arm and the S-LT arm must have 2 negative pregnancy tests before Lenalidomide treatment (Non-Childbearing potential: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy).
14. Participants with active hepatitis B Virus (HBV) are eligible if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 international units per milliliter (IU/mL); participants with untreated hepatitis C Virus (HCV) are eligible if viral load is negative per institutional standard; participants with human immunodeficiency virus (HIV) are eligible if cluster of differentiation 4 (CD4+) T-cell counts ≥350 cells per microliter (cells/μL), viral load is negative and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year.

Exclusion Criteria:

1. DLBCL with mucosa-associated lymphoid tissue (MALT) lymphoma; composite lymphoma (Hodgkin lymphoma + NHL); Gray zone lymphoma; DLBCL transformed from Chronic Lymphocytic Leukemia (Richter Syndrome); Primary mediastinal large B-cell lymphoma (PMBCL); T-cell rich large B-cell lymphoma.
2. Previous treatment with selinexor or other XPO1 inhibitors.
3. Contraindication to any drug contained in the different treatment arms.
4. Use of any standard or experimental anti-DLBCL therapy (including nonpalliative radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy) <21 days prior to Cycle 1 Day 1 (C1D1). Low dose steroids <30 mg prednisone (or equivalent) and palliative radiotherapy are permitted.
5. Received strong cytochrome P450 3A (CYP3A) inhibitors ≤7 days prior to Day 1 dosing or strong CYP3A inducers ≤14 days prior to Day 1 dosing.
6. Any AE, by Cycle 1 Day 1 (C1D1), which has not recovered to Grade ≤1 (CTCAE, v. 5.0), or returned to baseline, related to the previous DLBCL therapy, except alopecia.
7. Major surgery <14 days of C1D1.
8. Autologous stem cell transplant (SCT) <100 days or allogeneic SCT <180 days prior to C1D1 or active graft-versus-host disease after allogeneic SCT (or cannot discontinue graft versus host disease [GVHD] treatment or prophylaxis).
9. Prior chimeric antigen receptor T cell (CAR-T cell) infusion at any time (Phase 1 only); prior CAR-T cell infusion ≤120 days prior to C1D1 (Phase 2 only).
10. Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participant's safety, or able to comply with the study procedures.
11. Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
12. Inability to swallow tablets, malabsorption syndrome, or any other GI disease or dysfunction that could interfere with absorption of study treatment.
13. Breastfeeding women or pregnant women.
14. Inability or unwillingness to sign informed consent form.
15. In the opinion of the Investigator, participants who are below their ideal body weight and would be unduly impacted by changes in their weight.
16. Known allergy to any of the drug planned to be given.

    The following are Arm Specific exclusion criteria:
17. Arm B (S-PR): Serum total bilirubin >1.5 * ULN, Neuropathy Grade ≥2 (CTCAE, v5.0).
18. Arm C (S-PBR): Serum total bilirubin >1.5 * ULN, Neuropathy Grade ≥2 (CTCAE, v5.0).
19. Arm D (S-R-GemOx): Neuropathy Grade 2≥ (CTCAE, v5.0) interstitial lung disease or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) | Within the first cycle (maximum 28 days) of treatment
Phase 1: Recommended Phase 2 Dose (RP2D) | Up to 6 cycles (up to 6 months) of treatment
Phase 2: Overall Response Rate (ORR) per the Lugano Classification 2014 | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a complete response (CR) or partial response (PR) (up to 6 months)

SECONDARY OUTCOMES:
Phase 1: Overall Response Rate per the Lugano Classification 2014 | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a complete response (CR) or partial response (PR) (up to 6 months)
Phase 1: Disease Control Rate (DCR) per Lugano Classification 2014 | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a CR or PR or stable disease (SD) (up to 6 months)
Phase 1: Duration of Response (DOR) per Lugano Classification 2014 | Time from the first response of PR or CR until disease progression (up to 12 months)
Phase 1: Overall Response Rate (ORR) per the Modified Lugano Classification | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a CR or PR (up to 6 months)
Phase 1: Number of Participants With Adverse Events (AEs) by Occurrence, Nature, and Severity | From start of study drug administration up to 30 days after last dose of study treatment (up to 24 months)
Phase 2: Overall Response Rate per the Modified Lugano Classification | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a complete response (CR) or partial response (PR) (up to 6 months)
Phase 2: Disease Control Rate (DCR) per Lugano Classification 2014 | Cycle 1 Day 1 (each cycle consists of maximum 28 days) until a CR or PR or stable disease (SD) (up to 6 months)
Phase 2: Duration of Response (DOR) per Lugano Classification 2014 | Time from the first response of PR or CR until disease progression or death (up to 12 months)
Phase 2: Number of Participants With AEs by Occurrence, Nature, and Severity | From start of study drug administration up to 30 days after last dose of study treatment (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Arizona, Tucson, Arizona
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Irvine, Orange, California
  - US Oncology - Rocky Mountain Cancer Center, Aurora, Colorado
  - Loyola University Medical Center, Maywood, Illinois
  - Mission Cancer + Blood, Des Moines, Iowa
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - US Oncology - Oncology Associates of Oregon, Eugene, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - US Oncology - Prisma Health, Greenville, South Carolina
  - US Oncology - Texas Oncology Austin Midtown, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor Clinic - Mcnair Center, Houston, Texas
  - US Oncology - Northwest Cancer Specialists, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Undecided